CLINICAL TRIAL: NCT05579314
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Oral Dose Study to Assess Safety, Tolerability, Food Effect, Pharmacokinetics, and Pharmacodynamics of XW014 in Healthy Subjects and Patients With Type 2 Diabetes Mellitus
Brief Title: XW014 in Healthy Subjects and Patients With Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sciwind Biosciences USA Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: XW014-001
Record Dates: First submitted 2022-09-27; First posted 2022-10-13 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- SAD Cohort A - XW014 (Active Comparator): Single oral XW014 administration
  Interventions: Drug: XW014
- SAD Cohort A - Placebo (Placebo Comparator): Single oral placebo administration
  Interventions: Drug: Placebo
- MAD Cohort B - XW014 (Active Comparator): MAD in Healthy Subjects with Elevated BMI
  Interventions: Drug: XW014
- MAD Cohort B - Placebo (Placebo Comparator): MAD in Healthy Subjects with Elevated BMI
  Interventions: Drug: Placebo
- MAD Cohort C - XW014 (Active Comparator): MAD in Patients with T2DM
  Interventions: Drug: XW014
- MAD Cohort C - Placebo (Placebo Comparator): MAD in Patients with T2DM
  Interventions: Drug: Placebo
- MAD Cohort B-EXT - XW014 (Active Comparator): MAD in Healthy Subjects with Elevated BMI
  Interventions: Drug: XW014
- MAD Cohort B-EXT - Placebo (Active Comparator): MAD in Healthy Subjects with Elevated BMI
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XW014 — Oral tablets
  Arms: MAD Cohort B-EXT - XW014; MAD Cohort C - XW014
Drug: Placebo — Matched oral placebo tablets
  Arms: MAD Cohort B-EXT - Placebo; MAD Cohort C - Placebo
Drug: XW014 — Oral capsules
  Arms: MAD Cohort B - XW014; SAD Cohort A - XW014
Drug: Placebo — Matched oral placebo capsules
  Arms: MAD Cohort B - Placebo; SAD Cohort A - Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, first-in-human (FIH) study to evaluate the safety, tolerability, food effect (FE), pharmacokinetics (PK), and pharmacodynamics (PD) of orally administered XW014 in healthy participants and patients with T2DM. This study will consist of 4 parts: a Single Ascending Dose (SAD) part in healthy subjects (Part A), and Multiple Ascending Dose (MAD) parts in healthy subjects with elevated BMI (Part B and Part B-EXT) and patients with T2DM [Optional] (Part C).

DETAILED DESCRIPTION:
Part A - SAD, including FE cohort: Healthy participants with BMI in the range of ≥18.5 kg/m2 to ≤35.0 kg/m2 will be randomized to receive a single oral dose of either XW014 or placebo in each of the planned SAD cohorts.

Part B and Part B-EXT - MAD in healthy participants with elevated BMI: Healthy subjects with BMI in the range of ≥30 kg/m2 to ≤40.0 kg/m2 will be randomized to receive oral doses of XW014 or placebo in each of the planned MAD cohorts.

Part C - MAD in patients with T2DM: Patients with T2DM for at least 6 months, having hemoglobin A1c (HbA1c) in the range of 6.5% to 8.5% will be randomized to receive oral doses of XW014 or placebo in each of the planned MAD cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to participate in the study, give written informed consent, and comply with the study restrictions and all protocol procedures
2. Sex: male or female
3. Weight: >50 kg, inclusive, at screening
4. Age:

   1. For Part A 18 to 70 years, inclusive, at screening
   2. For Part B, Part B-EXT, and C 18 to 55 years, inclusive, at screening
5. Body Mass Index

   1. For Part A: ≥18.5 kg/m2 and ≤35.0 kg/m2, inclusive, at screening
   2. For Part B and Part B-EXT: ≥30.0 kg/m2 and ≤40.0 kg/m2, inclusive, at screening
   3. For Part C: ≥25.0 kg/m2 and ≤40.0 kg/m2, inclusive, at screening
6. Patients with T2DM for at least 6 months, having HbA1c of 6.5% to 8.5% (Part C)

Key Exclusion Criteria:

1. History or clinically significant active disease of the gastrointestinal, cardiovascular, hepatic, neurologic, renal, pancreatic, immunologic, dermatologic, endocrine, genitourinary, or hematologic system
2. Uncontrolled hypertension
3. History of type 1 diabetes mellitus
4. History or current diagnosis of acute or chronic pancreatitis or factors for pancreatitis
5. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2 or subjects with suspected medullary thyroid carcinoma
6. Existence of any surgical or medical condition that, in the judgment of the Investigator, might interfere with the absorption, distribution, metabolism, or excretion of the investigational product

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2024-11-16 (Actual); Study Completion 2024-11-16 (Actual)

PRIMARY OUTCOMES:
Number and percentage of treatment emergent adverse events (TEAE) and serious adverse events (SAE) | 11 weeks
Mean change from baseline in clinical laboratory values, vital signs, clinical findings from physical exam and ECG abnormalities | 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susan Xu, MD, Study Chair — Sciwind Biosciences
Locations (3):
- United States (3):
  - ICON - Early Development Services, Lenexa, Kansas
  - ICON - Early Development Services, San Antonio, Texas
  - ICON - Early Development Services, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No